CLINICAL TRIAL: NCT01506999
Title: GENOCOR Project-Laboratory of Genetic Mapping for Assessment of Cardiovascular Risk(GENOCOR LAB)
Brief Title: Genetic Mapping for Cardiac Risk Assessment
Acronym: GENOCOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Collaborators: Ministry of Education, Universities and Research, Italy (Other)
Responsible Party: Principal Investigator, Clara Carpeggiani, Senior Reasearcher of National research Council of Italy, Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Other Study IDs: GENOCOR
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Angina Pectoris; Myocardial Infarction; Coronary Disease; Myocardial Ischemia; Acute Coronary Syndrome
Keywords: Angina Pectoris; SNPs; Genetic; Myocardial Infarction; Cardiovascular Risk Factors
MeSH Terms: conditions — Angina Pectoris; Myocardial Infarction; Coronary Disease; Myocardial Ischemia; Acute Coronary Syndrome | interventions — Polymorphism, Single Nucleotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stable phase of ischemic heart disease: patients with history of angina pectoris, or myocardial infarction
  Interventions: Biological: MULTIGENE SCREENING FOR SINGLE SNPS
- acute phase of ischemic heart disease: patients with unstable angina or acute myocardial infarction
  Interventions: Biological: MULTIGENE SCREENING FOR SINGLE SNPS
- control group: subjects without ischemic heart disease (IHD)

INTERVENTIONS:
Biological: MULTIGENE SCREENING FOR SINGLE SNPS — DNA will be genotyped employing a multicolour assay system for SNPs based on TaqMan MGB (Minor Groove Binder) probes.
  Groups: Stable phase of ischemic heart disease; acute phase of ischemic heart disease

SUMMARY:
The main objective of the GENOCOR project (Genetic mapping for cardiac risk assessment) is the setting up of a joint public/private laboratory (GENOCOR-LAB) dedicated to the development and testing of new cost-effective technologies exploiting the growing knowledge in the genomic correlates of cardiovascular diseases (CVD) and of their evolution; the data obtained by the GENOCOR-Lab should especially orient secondary prevention and specific treatment of ischemic heart diseases (IHD).

DETAILED DESCRIPTION:
The Laboratory will be based in the premises of the CNR Institute of Clinical Physiology, a research institution operating as CVD Research Hospital System, with two Hospital Units (CNR Campus in Pisa and G. Pasquinucci Hospital in Massa).

The project is based on the cooperation of a national private company (DiaSorin, endowed with promising proprietary technologies in the novel diagnostic biotechnologies) and three research units (at clinical and molecular biology level) two from the National Research Council (IFC-CNR, Pisa and ITB-CNR, Milano, both very active in advanced biological research) and one from the University Vita-Salute San Raffaele (UHSR, Milano, operating a top range hospital and center for advanced biological research): GENOCOR Lab becomes then the first product of the cooperation within the CNR MERIT Network (MEdical Reseach in ITaly) currently being set-up by CNR.

The project is based on the availability of proprietary large scale databases of selected clinical populations that will be probed with the novel genomic and post-genomic technologies. High throughput SNPs technologies and post-genomic expression and proteomic analyses will be used to assess profiles of genetic variability identifying subjects with a distinct proneness to ischemic heart disease (IHD), hard cardiovascular events and unfavourable outcomes. Specific focusing will be made possible by the availability, within the proposed research network, of well established clinical data bases and biological sample collections, enabling the retrospective and prospective access to large and well characterised populations of patients with IHD. Cardiovascular phenotypes will include patients with acute coronary syndromes (unstable angina and acute myocardial infarction) and patients with chronic ischemic heart disease and prolonged follow-up; with this approach, it will be possible to cover both short-term and long-term evolution by detailed clinical, biohumoral and instrumental phenotyping at the time of acute events and with a systematic follow-up.

This approach should allow to overcome the major limitations and unbalance of previous studies, either focussed to small well characterized populations in which few genetic variations have been explored, or extended to large populations with a wider gene variability approach but inadequate information on phenotype and evolution disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by history of IHD with a non-fatal evolution(angina or AMI as first manifestation),age at the onset of the disease (<50 o >60 years.
* Patients with acute coronary syndrome as first manifestation of coronary disease, admitted to the coronary unit within 6 hours from the onset of symptoms.

Exclusion Criteria:

* Age>75
* Pregnancy
* Recent(< 6 months) cerebral ischemic attack
* Active cancer
* Inability to provide an informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by ischemic heart disease (IHD) with a non-fatal evolution. Patients with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2006-07; Study Completion 2012-07

PRIMARY OUTCOMES:
association studies between a panel of known SNPs of candidate genes and proneness to IHD and its prognosis; | 4 years
  High throughput SNPs technologies will be used to assess profiles of genetic variability identifying subjects with a distinct proneness to ischemic heart disease (IHD), hard cardiovascular events and unfavourable outcomes.
Number of participants with adverse events | maximum length of follow-up between enrollment and events or the planned end of follow-up
  Major cardiac and non-cardiac events will be register for the planned lenght of follow-up

SECONDARY OUTCOMES:
secondary prevention and specific treatment of ischemic heart diseases (IHD) | 10 years
  Understanding of genetic and molecular mechanisms of the different clinical syndromes of ischemic heart disease (IHD), of its patterns of evolution and response to treatment represents a key research issue to develop innovating approaches to early diagnosis, risk classification and treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CNR Institute of Clinical Physiology, Pisa, Italy

REFERENCES:
- [Derived] Carpeggiani C, Michelassi C, Landi P, L'Abbate A. Long-term prognosis of unheralded myocardial infarction vs chronic angina; role of sex and coronary atherosclerosis burden. BMC Cardiovasc Disord. 2018 Jul 31;18(1):156. doi: 10.1186/s12872-018-0890-5. PMID 30064378